CLINICAL TRIAL: NCT06565390
Title: Remote Oximeter Monitoring Post-discharge to Reduce Emergency Room Visits and Rehospitalization (ROMPER): A Randomized Clinical Trial
Brief Title: Remote Oximeter Monitoring Post-discharge to Reduce Emergency Room Visits and Rehospitalization
Acronym: ROMPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Owlet Baby Care, Inc. (Industry)
Responsible Party: Principal Investigator, Colm Travers, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 300013146; OSP 000545308 (Other Grant/Funding Number: Owlet Baby Care Inc.)
Record Dates: First submitted 2024-07-29; First posted 2024-08-22 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Intervention Model Description: The study will have two groups. One group will use the Owlet OSS 3.0 pulse oximeter and the other group will not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Babies in the Owlet monitor group (Experimental): The Owlet group will be given an Owlet OSS 3.0 monitor to wear when sleeping. The Owlet alarms if the baby has a very low heart rate or very low oxygen levels. In addition, caregivers in the Owlet group with a smart phone and Wi-Fi access will be able to use an application to monitor the baby's vital signs and sleep state. Will complete a survey or questionnaire every month until 6 months after discharge.
  Interventions: Device: Babies in the Owlet monitor group
- Babies in the Usual Care Group (No Intervention): The usual care group will not be given an Owlet vital sign monitor. Will complete a survey or questionnaire every month until 6 months after discharge.

INTERVENTIONS:
Device: Babies in the Owlet monitor group — The Owlet group will be given an Owlet OSS 3.0 monitor to wear when sleeping. The Owlet alarms if the baby has a very low heart rate or very low oxygen levels. In addition, caregivers in the Owlet group with a smart phone and Wi-Fi access will be able to use an application to monitor the baby's vital signs and sleep state.
  Arms: Babies in the Owlet monitor group

SUMMARY:
This randomized clinical trial will determine the efficacy of remote patient monitoring using an Owlet OSS 3.0 pulse oximeter for the reduction of emergency room visits and high-acuity rehospitalizations among high-risk infants after NICU discharge.

DETAILED DESCRIPTION:
To determine if among infants being discharged from the neonatal intensive care unit (NICU) without a cardiorespiratory monitor or respiratory support, remote patient monitoring using an Owlet OSS 3.0 pulse oximeter (Owlet, Lehi, UT) decreases emergency room visits and high-acuity rehospitalizations after discharge compared with routine care.

Infants being discharged from the neonatal intensive care unit (NICU) without a cardiorespiratory monitor or respiratory support are eligible for inclusion.

The Investigators will provide remote patient monitoring using an Owlet OSS 3.0 pulse oximeter to infants in the intervention group for a 6 month period. The Investigators will collect monthly outcome measures from caregivers of all infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants being discharged from the NICU
* Off all respiratory support (oxygen, CPAP, ventilator) before discharge home
* Gestational age ≥ 22 0/7 weeks' gestation at birth
* Parents/legal guardians have provided consent for enrollment

Exclusion Criteria:

* a major malformation, a neuromuscular condition that affects respiration or causes apnea, complex congenital heart disease and hemodynamically significant shunts, or terminal illness or decision to withhold or limit support.
* Infants being discharged from the neonatal intensive care unit (NICU) with a cardiorespiratory monitor or respiratory support are not eligible for inclusion.

Ages: 22 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 700 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Emergency room visits and high-acuity rehospitalizations. | 6 months
  Number of emergency room visits and high-acuity rehospitalizations.

SECONDARY OUTCOMES:
Number of participants with serious outcome events | 6 months
  The number of participants with serious adverse event composite outcome: includes death, medical provider delivered cardiac pulmonary resuscitation (CPR), receipt of positive airway pressure, or intubation during study period.
High-acuity rehospitalizations | 6 months
  The number of high-acuity rehospitalizations.
All-cause mortality. | 6 months
  The rate of all-cause mortality.
Other rehospitalizations | 6 months
  The number of other rehospitalizations.
Emergency room visits | 6 months
  The number of emergency room visits.
Sick visits | 6 months
  The number of sick visits mediated by wearing Owlet OSS 3.0 Sock while sleeping.
Apparent life-threatening event (ALTE/ Brief resolved unexplained event (BRUE) | 6 months
  Number of episodes of ALTE/BRUE
Healthcare utilization | 6 months
  Healthcare utilization in cost effectiveness analysis
Safe-sleep practice adherence | 6 months
  Number of participant caregivers reporting adherence to safe-sleep practices on questionnaire.
Caregiver sleep disturbance. | 6 months
  Caregiver sleep disturbance using the sleep quality scale.
Caregiver anxiety score. | 6 months
  Caregiver anxiety score assessed using State Trait Anxiety Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Colm P Travers, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
We will only share aggregate data with the study sponsor and with data analyst.